CLINICAL TRIAL: NCT06938607
Title: Post-operative Outcomes Comparing Drain vs No Drain Placement Following Anterior Cervical Discectomy and Fusion Surgery
Brief Title: Post-operative Outcomes of Anterior Cervical Discectomy and Fusion Surgery With and Without Drain Placement
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0199-25-FB
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: ACDF Surgery
Keywords: ACDF Surgery
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No-drain group: Participants assigned to the no-drain group will have their wound closed without a drain.
- Drain group: Participants assigned to the drain group will have a surgical drain placed on the surface of the wound during closure. The drain will be removed within 24 hours.
  Interventions: Device: Drain

INTERVENTIONS:
Device: Drain — Participants assigned to the drain group will have a surgical drain placed on the surface of the wound during closure. The drain will be removed within 24 hours.
  Groups: Drain group

SUMMARY:
Anterior Cervical Discectomy and Fusion (ACDF) is a widely performed surgical procedure used to treat cervical spondylosis and cervical disc herniations with cervical nerve root compression and or cervical spinal cord compression when conservative treatment options have been exhausted. The primary aim of ACDF is to alleviate neck, shoulder, and upper extremity pain associated with degenerative cervical disc disease by removing one or more affected discs, decompressing the nerves, and restoring cervical spine anatomy through the implantation of structural allograft/autograft bone or artificial spacers, plates, and screws. Historically, ACDF has demonstrated substantial long-term benefits in pain relief and quality of life improvements for patients. In the United States alone, the annual number of ACDF procedures exceeds 150,000 and is projected to rise significantly over the next four decades. Despite its technical complexity, ACDF is considered a relatively safe procedure. Common postoperative complications include dysphagia (1.7-9.5%), hematoma (0.4-5.6%), worsening myelopathy (0.2-3.3%), recurrent laryngeal nerve palsy (0.9-3.1%), cerebrospinal fluid leakage (0.5-1.7%), and surgical site infections (0.9-1.6%). One strategy employed to mitigate postoperative complications such as hematoma, surgical site infection, and the need for reoperation is the placement of an indwelling subfascial drain within the surgical site. These drains facilitate the removal of accumulated blood or serous fluid, thereby reducing localized pressure and potentially preventing adverse outcomes. Despite its theoretical benefits, the utility of subfascial drains remains a topic of debate among surgeons. Given the limited evidence on the efficacy of subfascial drain placement following ACDF, this study proposes a randomized controlled trial to evaluate the necessity and impact of subfascial drain placement on postoperative outcomes.

This study will determine whether subfascial drain placement reduces the incidence of postoperative complications, including hematoma, infection, airway compromise and secondary surgeries, compared to no drain placement following ACDF surgery; assess the impact of subfascial drain placement on the severity and duration of postoperative dysphagia compared to no drain placement; and evaluate participant-reported outcomes and satisfaction, including postoperative pain and recovery experience, between the drain and no-drain groups.

DETAILED DESCRIPTION:
Anterior Cervical Discectomy and Fusion (ACDF) is a widely performed surgical procedure used to treat cervical spondylosis and cervical disc herniations with cervical nerve root compression and or cervical spinal cord compression when conservative treatment options have been exhausted. The primary aim of ACDF is to alleviate neck, shoulder, and upper extremity pain associated with degenerative cervical disc disease by removing one or more affected discs, decompressing the nerves, and restoring cervical spine anatomy through the implantation of structural allograft/autograft bone or artificial spacers, plates, and screws. Historically, ACDF has demonstrated substantial long-term benefits in pain relief and quality of life improvements for patients. In the United States alone, the annual number of ACDF procedures exceeds 150,000 and is projected to rise significantly over the next four decades. Despite its technical complexity, ACDF is considered a relatively safe procedure. Common postoperative complications include dysphagia (1.7-9.5%), hematoma (0.4-5.6%), worsening myelopathy (0.2-3.3%), recurrent laryngeal nerve palsy (0.9-3.1%), cerebrospinal fluid leakage (0.5-1.7%), and surgical site infections (0.9-1.6%). One strategy employed to mitigate postoperative complications such as hematoma, surgical site infection, and the need for reoperation is the placement of an indwelling subfascial drain within the surgical site. These drains facilitate the removal of accumulated blood or serous fluid, thereby reducing localized pressure and potentially preventing adverse outcomes. Despite its theoretical benefits, the utility of subfascial drains remains a topic of debate among surgeons. Given the limited evidence on the efficacy of subfascial drain placement following ACDF, this study proposes a randomized controlled trial to evaluate the necessity and impact of subfascial drain placement on postoperative outcomes.

This study will determine whether subfascial drain placement reduces the incidence of postoperative complications, including hematoma, infection, airway compromise and secondary surgeries, compared to no drain placement following ACDF surgery; assess the impact of subfascial drain placement on the severity and duration of postoperative dysphagia compared to no drain placement; and evaluate participant-reported outcomes and satisfaction, including postoperative pain and recovery experience, between the drain and no-drain groups. Up to 360 participants will be randomly assigned to one of two groups. Those signed to the drain group will have a surgical drain placed on the surface of the wound during closure. The drain will be removed within 24 hours. Those in the no-drain group will have their wound closed without a drain. All other aspects of participants' care before and after surgery will be the same. No additional visits are required for this study. Basic information will be collected from participants' medical records, such as age, gender, type of surgery. For 180 days following surgery, participants' health will be monitored through clinical visit notes, phone calls with their doctor or clinic staff, and records of any hospital visits due to complications.

ELIGIBILITY:
Inclusion Criteria:

* 19-75 years of age
* Having elective anterior cervical discectomy and fusion (ACDF) surgery

Exclusion Criteria:

* Unable to stop anticoagulation medication
* Cervical (neck) cancer or tumor
* Combined anterior cervical discectomy and fusion, and posterior cervical fusion
* Active infection or trauma

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants scheduled to undergo a primary or revision single or multilevel anterior cervical discectomy and fusion (ACDF).
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Surgical Complications | Post-surgery 1-2 weeks, 3 months and 6 months
  Complications such as hematoma, infection, airway-compromise, and other complications will be recorded and monitored immediately after surgery and at followed-up visits, 1-2 weeks, 3 months and 6 months.

SECONDARY OUTCOMES:
Dysphagia Assessment EAT-10 | Post-surgery 1-2 weeks, 3 months and 6 months
  Dysphagia, the difficulty swallowing foods or liquids, will be assessed assessed at 1-2 weeks, 3 months and 6 months,using EAT-10 assessment tool. This tool has ten questions that are rated from 0 (no problem) to 4 (severe problem). Scores of 3 or above are considered abnormal.
Length of Hospital Stay | Post-surgery typically up to 1 week
  The total length of the post-surgical hospital stay will be obtained from medical records.
Post-operative Pain Assessment | Post-surgery 1-2 weeks, 3 months and 6 months
  Post-operative pain will be assessed using the self-reported numerical scale (0 - no pain, 10 - worst pain imaginable) at 1-2 weeks, 3 months and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cornett, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No